CLINICAL TRIAL: NCT05409937
Title: Influence of Wet Clothing on Thermal Protection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21-12H
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Low Body Temperatures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Improved Hot Weather Combat Uniform (Experimental): Wearing the Improved Hot Weather Combat Uniform; Asked to perform 60 min of standing with minimal movement, 60 min weighted (38.5lb) treadmill walking at 2.0mph, up to 4% grade, 60 min weight (38.5lb) treadmill walking at 2.5mph, up to 4% grade.
  Interventions: Other: Water-saturated Improved Hot Weather Combat Uniform
- Army Combat Uniform (Experimental): Wearing the Army Combat Uniform; Asked to perform 60 min of standing with minimal movement, 60 min weighted (38.5lb) treadmill walking at 2.0mph, up to 4% grade, 60 min weight (38.5lb) treadmill walking at 2.5mph, up to 4% grade.
  Interventions: Other: Water-saturated Army Combat Uniform
- Army Combat Uniform + Silk Weights (Experimental): Wearing the Army Combat Uniform + a base layer of silk weights; Asked to perform 60 min of standing with minimal movement, 60 min weighted (38.5lb) treadmill walking at 2.0mph, up to 4% grade, 60 min weight (38.5lb) treadmill walking at 2.5mph, up to 4% grade.
  Interventions: Other: Water-saturated Army Combat Uniform + Silk Weights
- Army Combat Uniform- XR (Experimental): Wearing the Army Combat Uniform; Asked to perform 60 min weighted (38.5lb) treadmill walking at 2.0mph, up to 4% grade, followed by 60 min of standing with minimal movement
  Interventions: Other: Water-saturated Army Combat Uniform

INTERVENTIONS:
Other: Water-saturated Improved Hot Weather Combat Uniform — Water-saturated Improved Hot Weather Combat Uniform
  Arms: Improved Hot Weather Combat Uniform
Other: Water-saturated Army Combat Uniform — Water-saturated Army Combat Uniform
  Arms: Army Combat Uniform; Army Combat Uniform- XR
Other: Water-saturated Army Combat Uniform + Silk Weights — Water-saturated Army Combat Uniform + Silk Weights
  Arms: Army Combat Uniform + Silk Weights

SUMMARY:
The aim of this investigation is to provide guidance for assessing the influence of wet clothing, and its drying time, on body temperature responses during cold air exposure. Twelve healthy and fit adults (men and women aged 18-49) will complete this study. Four cold air exposures (41°F, 180 min) will be randomly conducted, each while wearing a different clothing ensemble that has been saturated by water. During each cold air exposure, you will be asked to rest for 60 min and perform weighted (38.5lbs) treadmill walking for up to 120 min.

DETAILED DESCRIPTION:
Participants, in their first visit, will undergo baseline weighted treadmill walking consisting of ~20 min of treadmill walking with a load of 77lbs followed by ~25 min of treadmill walking with a load of 38.5lbs. They will also have their body composition evaluated (DEXA) and be fit for each uniform ensemble. This first laboratory visit will require ~3 hrs.

On separate days, participants will complete 4 experimental trials. After being submerged up to the neck in warm water for two minutes, three of the trials will ask that the participant move to a 41°F air environment, stand with minimal movement for 60 min, complete 60 min of weighted (38.5lb) treadmill walking at 2 mph, and up to 4% grade, and then complete 60 min of weighted (38.5lb) treadmill walking at 2.5 mph and up to 4% grade. Each of these three experimental trial visits will require ~5 hrs.

A single trial will ask that after being saturated in warm water, participants enter a 41°F air environment, immediately begin weighted treadmill walking (38.5lbs) at 2.0mph and up to 4% grade for a duration of 60 min before standing with minimal movement for 60 min. This trial will require ~4 hrs.

During all experimental trials, the primary outcomes include core temperature, measured continuously using a small pill inserted as a rectal suppository, and skin temperature, measured continuously using 11 small skin attached sensors. Secondary outcomes include metabolic rate, heart rate, thermal perceptions, and changes in body mass.

Non-federally employed civilians may be eligible to be paid $13.50/hour for participation (for a total of up to $310).

ELIGIBILITY:
Inclusion Criteria:

* Military or civilian, male or female, between the ages of 18 (17 if active duty military) and 49 years.
* Able to carry a rucksack weighing 35 kg (77lbs) for at least 20 minutes and able to carry a rucksack weighing 17.5kg (38.5lbs) for up to 120 minutes
* In good health as determined by our OMSO (Office of Medical Support and Oversight) General Medical Clearance.
* Vaccinated against COVID 19.
* Willing to refrain from heavy exercise and alcoholic beverages for 24 hours before each testing session.
* Willing to refrain from smoking or tobacco use for 8 hours before each testing session.
* Willing to refrain from caffeine ingestion for 12 hours before each testing session.
* Body fat percentage <18% for males, < 24% for females, once 6 individuals of higher body fat (18% or greater for males, 24% or greater for females) have completed the study.

Exclusion Criteria:

* History of cold injuries.
* Raynaud's syndrome.
* Cold-induced asthma/bronchospasm.
* Medications or dietary supplements that could alter cardiovascular, thermoregulatory, or vascular control.
* Heart, lung, kidney, muscle, or nerve disorder(s).
* Planned MRI during or within two days after completing the study.
* Known allergy to adhesives.
* Female and pregnant, planning to become pregnant, or breastfeeding.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Core Temperature | 5 hours
  Core temperature will be measured using a temperature pill that is inserted as a rectal suppository.
Skin Temperature | 5 hours
  Skin temperature will be measured using 11 different skin-attached temperature sensors.

SECONDARY OUTCOMES:
Heart Rate | 5 hours
  Heart Rate will be measured using telemetry [beats per min]
Oxygen Consumption/Metabolic Heat Production (MHP) | multiple 5 minute collections up to 1 hour
  Oxygen consumption and MHP will be assessed using computerized indirect calorimetry [ml/kg/min; Watts per meter squared]
Thermal Sensation (whole body, feet, and hands) | multiple 1 minute collections up to 1 hour
  Thermal sensation will be assessed using the American Society of Heating, Refrigerating and Air-conditioning Engineers Thermal Sensation Scale. This scale has numbers from -4 to +4 with every whole number accompanied by a verbal expression. The verbal expressions are used only to give the subject a relative feeling pertaining to the relative sensation. For example, -4 is associated with very cold whereas +4 is associated with very hot.
Thermal Comfort | multiple 1 minute collections up to 1 hour
  Thermal comfort will be assessed using a standard Thermal Comfort Scale. We will ask volunteers to rate how comfortable they feel with respect to temperature sensation. The scale has numbers ranging from 0 to 4 and with descriptors ranging from comfortable (0) to intolerable (4).
Perceived Skin Wetness | multiple 1 minute collections up to 1 hour
  Perceived Skin Wetness will be assessed using an adapted Skin Wetness Perception Scale. The scale ranges from 0 (extremely dry) to -6 (extremely wet; soaked).

CONTACTS AND LOCATIONS:
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seeley AD, Bodurtha PO, Greenfield AM, Pitsas DM, Shaw MA, Caldwell AR, Alba BK, Castellani JW, O'Brien C. Wet military uniforms pose low risk of hypothermia while static in mild cold air. Appl Physiol Nutr Metab. 2024 Dec 1;49(12):1763-1772. doi: 10.1139/apnm-2024-0180. Epub 2024 Sep 13. PMID 39270307